CLINICAL TRIAL: NCT04024553
Title: A Genetic Family Cohort Study of Bipolar Disorder in Chinese Han Population
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: CRC2018ZD02
Record Dates: First submitted 2019-06-12; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-06

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; family; genetic
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect 5 ml of venous blood of subjects with empty stomach into the 2% EDTA anticoagulation tube from 7 am to 9 am, for subsequent extraction of whole blood DNA and determination of plasma protein; simultaneously collect 2 ml of venous blood into PAXgene Blood RNA Tube and gently invert 10 times, placed vertically for subsequent extraction of whole blood RNA.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bipolar disorder family: Screening priori BD-I/BD-II patients， their relatives with mental illness (including but not limited to BD) and their healthy families.
- health control: Group-matched non-psychiatric family history health subjects were enrolled, DSM-IV-TR is used for demographic assessment.

SUMMARY:
This study intends to find out the pathogenic genes of bipolar disorder by collecting the two-phase family of Chinese Han population with the large sample using a family cohort study design, combined with the new generation of high-throughput sequencing technology and Genome-Wide Association Studies (GWAS), Proteomics, bioinformatics analysis, etc., which is expected to be clarified at the genetic level. The pathogenesis of bipolar disorder. At the same time, the investigators will conduct a five-year follow-up of cognitive function, brain function imaging and other major clinical symptoms in patients with bipolar disorder in the core family, and to explore familial bipolar disorder and sporadic biphasic. Differences in the clinical features of the disorder, in order to explore sensitive and specific biomarkers from a multidimensional perspective (cognitive function, brain imaging, genetic features, clinical features, etc.), which may contribute to bipolar disorder in the future. Accurate diagnosis and early identification and prevention have important scientific significance and clinical diagnosis and treatment significance.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a serious, complex, family-grafting mental illness. Studies have shown that genetic factors may be the dominant factor in the pathogenesis of bipolar disorder, thus, it is worth looking forward to getting started and clarifying the etiology of bipolar disorder from a genetic perspective. However, earlier genetic studies such as linkage analysis, genetic mutation detection (preferred candidate genes), and recent genetic studies (no need to presuppose candidate genes) such as Whole Genome Sequencing (WGS), whole genome GWAS and Whole-exome sequencing (WES) failed to identify any biogenic disorder gene or chromosomal region that plays a major role in, which may be related to the synergy of population heterogeneity, insufficient sample size or coordination effect caused by common mutations.

As a familial, highly heritable psychiatric disease, the literature suggests that the pathogenic genes of bipolar disorder may be directly derived from the intergenerational transmission of rare mutations in family members, and these rare variants are more likely to be predicated from the family. It has been found that the family has a higher frequency and is more susceptible to detecting susceptibility genes for bipolar disorder. Therefore, the family research design combined with WGS, GWAS and other advanced genetic research methods can reduce the unnecessary sample size, eliminate the confounding factors of the population, and more easily capture the potential genes of bipolar disorder.

However, at present, there are few reports of foreign bipolar disorder family and the results are not consistent. There is no research report on the large sample family of Chinese Han population in China. Therefore, it is necessary to expand the family sample size and combine with new genetic research methods in the Han population. explore. Therefore, this study intends to find out the pathogenic genes of bipolar disorder by collecting the two-phase family of Chinese Han population with the large sample using a family cohort study design, combined with the new generation of high-throughput sequencing technology and GWAS, Proteomics, bioinformatics analysis, etc., which is expected to be clarified at the genetic level. The pathogenesis of bipolar disorder. At the same time, the investigators will conduct a five-year follow-up of cognitive function, brain function imaging and other major clinical symptoms in patients with bipolar disorder in the core family, and to explore familial bipolar disorder and sporadic biphasic. Differences in the clinical features of the disorder, in order to explore sensitive and specific biomarkers from a multidimensional perspective (cognitive function, brain imaging, genetic features, clinical features, etc.), which may contribute to bipolar disorder in the future. Accurate diagnosis and early identification and prevention have important scientific significance and clinical diagnosis and treatment significance.

ELIGIBILITY:
Inclusion Criteria:

* BD patients from BD family:

  1. Meets the diagnostic criteria of BD in DSM-IV-TR, does not limit subtypes and current disease status;
  2. age ≥ 15 years old;
  3. Han nationality;
  4. There are enough audition levels to complete the necessary examinations for the study;
  5. Understand the research content and sign the informed consent form. If the patient is unable to sign the informed consent form due to the young age, senior age, low education level or other reasons, they can be signed by their relatives or signed by their guardian.
* Healthy menbers from BD family:

  1. age ≥ 15 years old;
  2. Han nationality;
  3. biological parents or compatriots of the proband, cousins;
  4. There are enough audition levels to complete the necessary examinations for the study;
  5. Understand the research content and sign the informed consent form. If the patient is unable to sign the informed consent form due to the young age, senior age, low education level or other reasons, they can be signed by their relatives or signed by their guardian.
* Healthy control enrollment criteria without family history:

  1. age ≥ 15 years old;
  2. Han nationality;
  3. gender matches the patient group in the family;
  4. There are enough audition levels to complete the necessary examinations for the study;
  5. Understand the research content and sign the informed consent form. If the patient is unable to sign the informed consent form due to his or her age, advanced age, low education level or other reasons, he or she may be entrusted to sign by his or her relatives or signed by his guardian;

Exclusion Criteria:

* BD patients from BD family:

  1. There is a DSM-IV-TR axis II disease (mental retardation, etc.) that significantly affects the patient's current state of mind;
  2. There are serious physical diseases, it is difficult to complete the necessary examinations, including history of brain trauma or cerebrovascular disease, severe cirrhosis, acute and chronic failure, severe diabetes, aplastic anemia, moderate to severe malnutrition and other serious nerves, heart, Physical diseases such as liver, kidney, endocrine, and blood system or diseases that may interfere with the test evaluation (the abnormal index is more than 2 times higher than the normal value).
* Healthy menbers from BD family and healthy control enrollment criteria without family history::

  1. with a mental disorder that meets the diagnostic criteria for DSM-IV-TR axis I or who have suspected psychosis but do not meet the diagnostic criteria;
  2. There are DSM-IV-TR axis II diseases (mental retardation, etc.) that significantly affect the patient's current mental state;
  3. There are serious physical illnesses, and it is difficult to complete the necessary examinations.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We intend to expand the sample size of the family, and collect 50 core families and 200 healthy controls at this stage. Similarly, during the validation phase, it is proposed to include 30 core families for verification.
  To verify the results of the first part of the study in sporadic BD patients and healthy controls, 783 patients with sporadic BD and 692 healthy controls were calculated by sample size estimation formula. With drop-off rate of 20%, 939 cases and 830 cases are needed respectively. In order to avoid other factors falling off, it is proposed to include 1000 cases of sporadic BD patients and healthy controls respectively.
Sampling Method: Probability Sample
Enrollment: 2520 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Potential risk genes | at december 2022
  The investigators will collect peripheral blood samples of patients and healthy controls during the baseline period, and blood samples from family members during follow-up period. The blood will be used for WGS, GWAS, WES to get candidate genes. Reported high risk genes such as CACNA1C、DTNA、FOXP1 and so on are the focus.

SECONDARY OUTCOMES:
HAMD-17 scores of patients and high-risk subjects | by december 2022
  Hamilton depression scale is used to assess subjects at the baseline and every follow-up point(health controls are assessed only at baseline). HAMD is the most commonly used scale for clinically assessed depression. Total score < 7 points means normal; total scores in 7~17 points indicates that there may be depression; total scores in 17~24 points shows that there must be depression; total score >24 points means major depression.
Onset age of BD subjects | by december 2022
  Data of onset age will be record since the subjects join this peoject, and the invetigators will continue recording especially at each follow-up point.
Wisconsin Card Sorting Test results | by december 2022
  The family members will be tested at baseline and 5 follow-up periods, totally 6 times. The healthy control will be tested once at baseline. Wisconsin Card Sorting Test (WCST) reflects congnitive function, which includes 13 indexes. Higher scores indicate better congnition.
Characteristic changes of electroencephalogram | by december 2022
  In this study the investigators use EEG equipment from BrainProducts of Germany. The sampling frequency is 1000hz. Detection items include gamma resonance, mismatched negative wave MMN, auditory event related potential P300, visual event related potential P300, and resting EEG. Family members were tested for the baseline period and subsequent annual follow-up period, a total of 6 times. Healthy controls test once at the baseline period.
YMRS scores of patients and high-risk subjects | by december 2022
  Young's Mania Rating Scale is used to assess subjects at the baseline and every follow-up point(health controls are assessed only at baseline). It is mainly used to assess the symptoms and severity of mania, which includes 11 items. Total scores range from 0 to 60, higher scores means the symptoms are more severe.
Course of disease of BD subjects | by december 2022
  Disease course will be record since the subjects join this peoject, and until the end of this study.
Treatment plan of BD subjects | by december 2022
  Treatment of BD patients will be record since the subjects join this peoject, and the invetigators will continue recording especially at each follow-up point.
STROOP test results | by december 2022
  The family members will be tested at baseline and 5 follow-up periods, totally 6 times. The healthy control will be tested once at baseline. STROOP test is a Cognitive psychology test, which is also called color word conflict test. In the randomly appearing text combinations, subjects are supposed to quickly read out names of colors according to the color of the text, and then the reading time is compared in this study.
Repetitive Neuropsychological Status test (RBANS) results | by december 2022
  The family members will be tested at baseline and 5 follow-up periods, totally 6 times. The healthy control will be tested once at baseline. RBANS is a test for subjects' neuropsychological state. It has 12 tasks. The original score will be converted to a standard score with a total score of 100 points. Higher scores means better congnitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, Principal Investigator — Shanghai Mentao Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China